CLINICAL TRIAL: NCT04318496
Title: Acupuncture for Blunt Chest Trauma: A Protocol for a Double-Blind Randomized Control Trial
Brief Title: Acupuncture for Blunt Chest Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Peiyu Kao, Principal Investigator, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH109-REC1-002
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Chest Trauma; Rib Fractures
Keywords: Blunt chest trauma; Acupuncture; Press tack needle; Rib fracture
MeSH Terms: conditions — Thoracic Injuries; Rib Fractures

STUDY DESIGN:
Intervention Model Description: Double Blinded Randomized Control Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study nurse 1 will be responsible to randomize and prepare the needles in the envelopes. Outside the envelopes, there will be a number belonged to one patient, and inside the envelopes, there will 14 separate sterile needle which can be either placebo or true press tack needles. The envelopes and the pouches of needle will look the same. The acupuncturist will be asked not to check the needles when they insert them. At the time of acupuncture, a nurse will accompany the acupuncturist and will verify that he is not examining the needles closely. Study nurse 2 will do the measurement. The acupuncturist, patients and study nurse 2 will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture with press tack needle group (Acu) (Experimental): the press tack needles (PYONEX Φ0.20×0.6 mm made by Seirin Corporation) has a diameter of 0.2 mm and length of 0.6 mm will be used on the following bilateral points; GB 36 (Waiqiu), GB 34 (YangLingQuan), ST 36 (Zusanli), LI 4 (HeGu), LU 7 (LieQue), TH 5 (Waiguan) press tack needles retention time will be 4 days.
  Interventions: Other: Press Tack Acupuncture
- Placebo group (Con) (Placebo Comparator): The pess tack placebo is PYONEX sticker and pack that is identical to the press needle, except that the needle part was removed. The acupuncturist will apply the stickers on the following bilateral acupoints: GB 36 (Waiqiu), GB 34 (YangLingQuan), ST 36 (Zusanli), LI 4 (HeGu), LU 7 (LieQue), TH 5 (Waiguan) press tack stickers retention time will be 4 days.
  Interventions: Other: Press Tack Placebo

INTERVENTIONS:
Other: Press Tack Acupuncture — PYONEX Φ0.20×0.6 mm made by Seirin Corporation
  Other Names: Press Tack Needle/ sticker needle/ PYONEX
  Arms: Acupuncture with press tack needle group (Acu)
Other: Press Tack Placebo — PYONEX placebo sticker made by Seirin Corporation
  Other Names: PYONEX placebo
  Arms: Placebo group (Con)

SUMMARY:
Introduction:

Chest blunt trauma accounts in up to 65% of polytrauma patients. In patients with 0-2 rib fracture, the treatment is relatively limited to oral pain killer and breathing exercise. The patients will suffer two weeks of severe pain accompanied with poor sleep and inability to preform simple daily live activities. In this double blind randomized control study, the investigators offer acupuncture as an additional treatment option.

Methods:

The study is a double blind randomized control trial. the study will include the press needle acupuncture (Acu) and placebo (Con) group. Both groups will receive one treatment, following the first visit to the clinic after chest trauma accident.

DETAILED DESCRIPTION:
Introduction:

Chest blunt trauma accounts in up to 65% of polytrauma patients. In patients with 0-2 rib fracture, the treatment is relatively limited to oral pain killer and breathing exercise. The patients will suffer two weeks of severe pain accompanied with poor sleep and inability to preform simple daily live activities. In this double blind randomized control study, the investigators offer acupuncture as an additional treatment option.

Methods:

The study is a double blind randomized control trial. the study goal is to examine the effect of acupuncture on patients with chest trauma. the study will include totally 72 patients and divide them to two group; the press needle acupuncture (Acu) and placebo (Con) group. Both groups will receive one treatment, following the first visit to the clinic after chest trauma accident. Follow up time will be 3 months.

Expected outcome:

The results of this study can potentially provide a simple and cost effective provide analgesic solution to blunt chest trauma patients. The study design can serve as supporting evidence for future double blind studies in acupuncture.

Other information:

The study will be conducted in thoracic surgical department and acupuncture department in China medical university hospital, Taichung, Taiwan. The study is conducted on blunt chest injury patients and is anticipated to have minimum risk for adverse events. Enrollment of the patients and data collection will start after March 2020. The study expected completion time will be March 2022.

Keywords: blunt chest trauma, acupuncture, press tack needle, rib fracture

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 year-old
* Patients have chest trauma described by themselves or medical chart record within one week
* Injury Severity Score (ISS) is less than 18 points
* Body Mass Index(BMI)<30

Exclusion Criteria:

* Sternal fracture
* Injury Severity Score (ISS) is equal or more than 18 points
* History of intercostal nerve injury
* History of cardiovascular disease
* History of chronic lung disease
* Significant lung mass or chest deformity noted in the chest plain film

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) - rest | 3 months
  pain scale form 1-10 when 10 is the most painful
Numerical Rating Scale (NRS) - mobile | 3 months
  pain scale form 1-10 when 10 is the most painful

SECONDARY OUTCOMES:
Visual Analogue Pain Scale (VAS) | 4 days
  Pain scale form 1-10 when 10 is the most painful
Face Rating Scale (FRS) | 4 days
  Face expression pain scale. scores form 0-5 when 5 is the most painful
Flow meter | 4 days
  Measure the amount of air the patient can exhale, It has three chambers with their own balls that requires air pressures from 600-1200 cc per second. 1200cc is the highest score and indicates good exhalation
Verran and Snyder-Halpern sleep scale | 4 days
  includes 15 question on the patients sleep quality, each question has a 100mm line. Patients will raking each question 0-100 when 100 means no existing insomnia
Chest plain film | 4 days
  Chest X-ray, will help examine the number of rib fractures, the incidence of hemothorax and pneumothorax
Pain killer or muscle relaxant medication does used | 4 days
  We will measure the amount of analgesic or muscle relaxant medication each patient used

CONTACTS AND LOCATIONS:
Overall Officials: Peiyu Kao, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- Out-Patient Clinic of China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kao PY, Lottering B, Lu TY, Ho WC, Lin YS, Huang TM, Chen CK, Chen JX, Lee YC, Chen FP, Ben-Arie E. Press tack needle stimulation for blunt chest trauma: a randomized double-blind control trial. Interact Cardiovasc Thorac Surg. 2022 Jun 15;35(1):ivac158. doi: 10.1093/icvts/ivac158. PMID 35670748
- [Derived] Kao PY, Ben-Arie E, Lu TY, Ho WC, Lee YC, Lin YS, Chen CK, Chen JX, Huang TM, Chen FP. Acupuncture for blunt chest trauma: A protocol for a double-blind randomized control trial. Medicine (Baltimore). 2021 May 7;100(18):e25667. doi: 10.1097/MD.0000000000025667. PMID 33950945